CLINICAL TRIAL: NCT05169528
Title: Colorectal Cancer Prehabilitation in Changi General Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Kwok Kah Meng, Consultant, Changi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIRB Ref No.:2020/2063
Record Dates: First submitted 2021-11-30; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal; Cancer Prehabilitation; Novel; Model of Care
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: before-after trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal Cancer Prehabilitation Program (Other): This is a before-after trial. The same group of participants will have a series of outcome measures taken at baseline, which will then be compared to these same outcome measures when repeated after undergoing prehabilitation and at 3 months' post-operatively
  Interventions: Other: Colorectal Cancer Prehabilitation Programme

INTERVENTIONS:
Other: Colorectal Cancer Prehabilitation Programme — Assessment and Interventions involving the Prehabilitative domains of medical optimisation, exercise prescription, nutrition and mental health optimisation

SUMMARY:
Cancer prehabilitation typically involves multiple pre-op visits. The investigators aim to assess the impact of their novel model, a "one-stop "service by a small, "levelled-up" core team on newly diagnosed colorectal cancer patients planned for surgery.

DETAILED DESCRIPTION:
Objective Cancer prehabilitation typically involves multiple pre-op visits. The investigators aim to assess the impact of their novel model, a "one-stop "service by a small, "levelled-up" core team on newly diagnosed colorectal cancer patients planned for surgery.

Design This is a before-after trial in a tertiary public hospital in Singapore, involving all newly diagnosed colorectal cancer patients planned for surgery who are referred to the Cancer Prehabilitation Program. The primary outcome measure is the 6-minute-walk-test. Others include physical, psychological, quality-of-life and post-operative measures, and patient-satisfaction-surveys, taken at baseline, pre-operatively (post-prehabilitation), and 3-months-post-operatively.

Keywords: Colorectal; Cancer Prehabilitation; Novel; Model of Care

ELIGIBILITY:
Inclusion Criteria:

1. All newly diagnosed colorectal cancer patients planned for surgery in Changi General Hospital, Singapore

Exclusion Criteria:

1. Patients' refusal to participate

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
6-minute-walk-test | Baseline
  Distance walked in 6 minutes under standardised conditions
6-minute-walk-test | Pre-Operatively (after prehabilitation)
  Distance walked in 6 minutes under standardised conditions
6-minute-walk-test | Post-Operatively (3 months)
  Distance walked in 6 minutes under standardised conditions

SECONDARY OUTCOMES:
30-second-sit-to-stand-test | Baseline
  Number of repetitions of sit-to-stand within 30 seconds
30-second-sit-to-stand-test | Pre-Operatively (after prehabilitation)
  Number of repetitions of sit-to-stand within 30 seconds
30-second-sit-to-stand-test | Post-Operatively (3 months)
  Number of repetitions of sit-to-stand within 30 seconds
Hospital Anxiety and Depression Scale | Baseline
  Divided into Anxiety (0-21 points) and Depression scale (0-21 points), the higher the worser
Hospital Anxiety and Depression Scale | Pre-Operatively (after prehabilitation)
  Divided into Anxiety (0-21 points) and Depression scale (0-21 points), the higher the worser
Hospital Anxiety and Depression Scale | Post-Operatively (3 months)
  Divided into Anxiety (0-21 points) and Depression scale (0-21 points), the higher the worser
EuroQol- 5 Dimension | Baseline
  Health Score (visual analogue scale from 0-100), the higher the better
EuroQol- 5 Dimension | Post-Operatively (3 months)
  Health Score (visual analogue scale from 0-100), the higher the better
Post-Operative Hospital Length of Stay | From Date of Admission for Surgery till Date of Discharge, assessed up to 100 weeks
  Post-Operative Hospital Length of Stay
30-Day Post-Operative Major Complications | From Surgery till 30 Days Post-op
  30-Day Post-Operative Major Complications
30-Day Post-Operative Readmission Rates | From Surgery till 30 Days Post-op
  30-Day Post-Operative Readmission Rates
30-Day Post-Operative Mortality | From Surgery till 30 Days Post-op
  30-Day Post-Operative Mortality
Patient Satisfaction Survey | Pre-Operatively (after prehabilitation)
  Patient Satisfaction Survey
Patient Satisfaction Survey | Post-Operatively (3 months)
  Patient Satisfaction Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No